CLINICAL TRIAL: NCT05720611
Title: Growing Health Hearts: An Online Gardening Program for Adults With Risk Factors for Cardiovascular Disease
Brief Title: Growing Healthy Hearts: An Online Gardening Program for Adults With Risk Factors for Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Susan Veldheer, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00017020
Record Dates: First submitted 2023-01-13; First posted 2023-02-09 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group will consist of a digitally delivered course designed to teach gardening, cooking and nutrition education to adults with risk factors for CVD. Participants will be invited to participate in 10 Zoom-based gardening and cooking education sessions. Zoom meetings will be facilitated by members of the study team, will present information to participants and will allow participants to ask questions and share their experiences with others. The materials will walk the participant through various aspects of starting and tending a garden. Participants will be asked to engage in a closed Facebook group.
  Interventions: Behavioral: Digitally delivered gardening and healthy eating course
- Control Group (Placebo Comparator): Participants in this group will complete all questionnaires but will not receive the digitally delivered course or access to Facebook.
  Interventions: Behavioral: Digitally delivered gardening and healthy eating course

INTERVENTIONS:
Behavioral: Digitally delivered gardening and healthy eating course — The intervention group will consist of a digitally delivered course designed to teach gardening, cooking and nutrition education to adults with risk factors for CVD. Participants will be invited to participate in 10 Zoom-based gardening and cooking education sessions. Zoom meetings will be facilitated by members of the study team, will present information to participants and will allow participants to ask questions and share their experiences with others. The materials will walk the participant through various aspects of starting and tending a garden.

SUMMARY:
This study aims to assess the effectiveness on an online gardening study for beginner gardeners with the goal of improving diet and physical activity in those with at least one risk factor for cardiovascular disease.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility of an online gardening and nutrition intervention in adults with risk factors for cardiovascular disease using a randomized controlled trial design. During the trial, the intervention condition will learn how to start a garden plot (either at home or in a community garden) and grow fruits and vegetables for personal consumption. We will also provide this group with nutrition education related to the DASH diet and basic cooking skills instruction. The control condition participants will receive no intervention during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 20 years old
2. Have any one or more health condition(s) or risk factor(s) for CVD. These include, but are not limited to:

   1. Any history of cardiovascular disease
   2. Any family history of cardiovascular disease (as measured by asking if both living and deceased, close biological relatives, that is, blood relatives including father, mother, sisters or brothers, ever told by a health professional that they had a heart attack or angina before the age of 50)
   3. Any history of stroke or DVT
   4. High cholesterol
   5. High blood pressure
   6. Overweight/obesity (BMI >=25)
   7. Diabetes, prediabetes, or borderline diabetes
   8. Current or past Tobacco use
3. Reports consuming fruit and vegetables less than 5 times per day
4. Report less than 150 minutes of physical activity per week
5. Have access to stable and consistent internet access
6. Have a Facebook account or willing to open a Facebook account
7. Have a smart phone or computer and capacity to download the Fitbit app or Fitbit Connect Software
8. Must be willing to wear a Fitbit tracker almost continually (23.5 hours/day) for duration of study
9. Have access to a kitchen in or near their living space
10. Has access to space to start a garden (at home or in a community garden either in the ground, raised beds, or containers)

Exclusion Criteria:

1. Unwilling to participate in Zoom sessions and have their voice and face recorded for research purposes.
2. Currently tends a vegetable garden (as measured by if they have tended a garden in the past year or are planning to tend a garden (outside of this study) in the coming season)
3. Moving out of the area in the next 5 months
4. Non-English speaking or reading
5. Pregnant women
6. Participation in a past FCM gardening intervention study
7. Medical conditions or medications that limit ability to freely increase dietary intake of fruits and vegetables (e.g., kidney failure, dialysis)
8. A medical condition that precludes safe pursuit of gardening, i.e., recent heart conditions (e.g., heart failure, stroke, heart attack), recent or pending surgery, severe orthopedic conditions, pending hip/knee replacement, paralysis, dementia, unstable angina or uncontrolled arrhythmias, or uncontrolled asthma or allergies.
9. Close contacts of current participants in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Acceptability | 24 weeks
  Participant acceptability of the program based on 80% of intervention participants providing an average rating of the intervention as 4 or higher on the Weiner Acceptability Scale

SECONDARY OUTCOMES:
Demand | Baseline and 24 weeks
  Participant demand in terms of 1) ability to recruit 40 participants at baseline and 2) ability to retain at least 70% of participants as measured by number of participants who complete the follow up questionnaires at the 24 week time point
Practicality | 24 weeks
  80% of intervention group participants report completing 16 out of 20 gardening-related study tasks.
Fruit and vegetable intake | From baseline to 24 weeks
  Between group differences in servings of fruits and vegetables from baseline to 24 weeks as assessed by the National Cancer Institute's Diet History Questionnaire 3
Physical activity | From baseline to 24 weeks
  Between group differences in minutes of self-reported physical activity from baseline to 24 weeks as assessed by the International Physical Activity Questionnaire short form.
Cooking confidence | From baseline to 24 weeks
  Between group differences in self-reported cooking confidence score as assessed by the Cooking and Food Skills (Lavelle et al. 2017)
Gardening confidence | From baseline to 24 weeks
  Between group differences in total gardening confidence score as assessed by a 20 item gardening task questionnaire on confidence to complete gardening tasks using a 10 point Likert scale.
Gardening enjoyment | From baseline to 24 weeks
  Between group differences in the total intrinsic motivation score for gardening activity as measured by the Intrinsic Motivations Questionnaire.
Social support-Healthy eating | From baseline to 24 weeks
  Between group differences the self-reported Social Support for Healthy Eating Questionnaire (Salis et al., 1987).
Social support-physical activity | From baseline to 24 weeks
  Between group differences in the self-reported Social Support for Physical Activity Questionnaire (Salis et al, 1987)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Veldheer S, Rutt K, Schaefer E, Kim I, Hrabovsky S, Smith B, Thomas OW, Moore AM, Pagoto S, Conroy DE, Schmitz KH, Sciamanna C. Growing Healthy Hearts: a pilot randomized controlled trial of a digitally delivered gardening, cooking, and Dietary Approaches to Stop Hypertension (DASH) diet intervention for adults with cardiovascular risk factors. Pilot Feasibility Stud. 2026 Jan 28. doi: 10.1186/s40814-026-01766-1. Online ahead of print. PMID 41606653